CLINICAL TRIAL: NCT00892333
Title: Repair of Large Abdominal Hernia Defects By A Novel Biologic Mesh: A Prospective Multi-Center Observational Study
Brief Title: Large Abdominal Hernia Repair With SurgiMend 3.0
Acronym: BRIDGE
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Massachusetts General Hospital (Other); Boston Medical Center (Other); Cook County Hospital (Other); University of Southern California (Other); Yale University (Other); Oregon Health and Science University (Other); State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: TEI-002
Record Dates: First submitted 2009-04-29; First posted 2009-05-04 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Hernia
Keywords: Repair of a large hernia with SurgiMend 3.0, a biologic mesh
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The rate of hernia recurrence at one year following repair of a large abdominal hernia with a biologic mesh is high, ranging from 30% to 100%, with a reported historic average rate of 40%. The purpose of this study is to evaluate the rate of hernia recurrence at one year following repair with SurgiMend 3.0, an FDA-cleared novel biologic mesh, the hypothesis being that such rate will be less than 20% at one year, representing a 50% reduction over the historic rate of 40%.

ELIGIBILITY:
Inclusion Criteria:

All three of the following criteria must be present for enrollment into the study:

* Large abdominal hernia
* Inability to close the fascia primarily
* Contra-indication for the use of synthetic mesh
* Age > 18 years

Exclusion Criteria:

* Use of SurgiMend 3.0 to simply reinforce a complete closure of the fascia performed either primarily or sequentially or by component separation technique
* Inability to close the skin over the SurgiMend 3.0

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with surgical conditions such as i) open abdomen after a damage control operation for a traumatic or non-traumatic surgical emergency, ii) removal of infected prosthetic materials from a previous abdominal hernia repair, iii) iatrogenic injury of the bowel during adhisiolysis for repair of a large abdominal hernia, iv) contaminated operative field due to presence of an ostomy or the need for additional surgical procedures.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2009-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George C Velmahos, MD, Ph.D., Principal Investigator — Massachusetts General Hospital/ Harvard University
Locations (8):
- United States (8):
  - Los Angeles County/University of Southern California Medical Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Cook County Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - State University of New York (SUNY), Upstate Medical Center, Syracuse, New York
  - Oklahoma University, Oklahoma City, Oklahoma
  - Oregon Health and Science University (OHSU), Portland, Oregon